CLINICAL TRIAL: NCT00673257
Title: Pharmacokinetics of Daunomycin in Children
Brief Title: Pharmacokinetics of Daunorubicin in Young Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ABTR06C1; CDR0000490024 (Other: Clinical Trials.gov); COG-ABTR06C1 (Other: Children's Oncology Group); NCI-2009-00327 (Other: Registry ID: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-02

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pharmacokinetics of Daunorubicin chemotherapy patients (Experimental): Patients receiving a chemotherapy regimen including daunorubicin hydrochloride administered as an infusion of any duration < 24 hours on a 1 or a 2 day schedule. Pre-study evaluations no greater than 14 days prior to daunomycin administration. If patients have had significant intercurrent illness or treatment that might affect organ function, laboratory work should be performed at an appropriately closer interval to daunomycin administration. A complete history and physical examination including height, weight and body surface area. Patients should be weighed with only light clothing; shoes must be removed before weight is measured. Patients height should be measured using a stadiometer after removing shoes. Laboratory evaluation: a) CBC with differential and platelet count. b) ALT, AST, bilirubin, creatinine, total protein, albumin, alkaline phosphatase, GGT.
  Interventions: Other: pharmacological study; Procedure: dual x-ray absorptimetry

INTERVENTIONS:
Other: pharmacological study — pharmacological studies
Procedure: dual x-ray absorptimetry
  Other Names: DEXA scan; dual energy x-ray absorptimetry

SUMMARY:
This laboratory study is looking at the pharmacokinetics of daunorubicin in young patients with cancer. Collecting and storing samples of blood from patients with cancer to study in the laboratory may help doctors learn more about how patients respond to treatment with certain chemotherapy drugs.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pharmacokinetics of daunorubicin hydrochloride in pediatric patients with malignancy.

Secondary

* Evaluate the relationship between body composition (percent body fat) and the pharmacokinetics of daunorubicin hydrochloride in these patients.
* Correlate the pharmacokinetics of daunorubicin hydrochloride with gender, age, or ethnic background in these patients.
* Explore, in a preliminary fashion, possible relationships between pharmacokinetic results and toxicity.
* Explore, in a preliminary fashion, possible relationships between pharmacokinetic results and renal and hepatic function and complete blood count.
* Explore, in a preliminary fashion, possible genetic polymorphisms that may influence daunorubicin hydrochloride disposition.

OUTLINE: This is a multicenter study.

Patients undergo blood collection prior to, periodically during, and after treatment with daunorubicin hydrochloride for pharmacokinetic analysis.

Patients also undergo body composition testing within 7 days before or after the administration of daunorubicin hydrochloride using dual-energy x-ray absorptiometry.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any malignancy
* Must be receiving a chemotherapy regimen that includes daunorubicin hydrochloride administered as an infusion of any duration for < 24 hours on either a 1- or a 2-day schedule, including bolus and all short infusion schedules

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* No significant uncontrolled systemic illness
* Large implanted prostheses allowed (should not undergo dual energy x-ray absorptiometry scan)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2007-01; Primary Completion 2011-07 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey L. Berg, MD, Study Chair — Texas Children's Cancer Center
Locations (60):
- United States (56):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- Swiss Pediatric Oncology Group Bern, Bern, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pharmacokinetics of Daunorubicin Chemotherapy Patients
Started | 107
Completed | 102
Not Completed | 5
Not completed — Withdrawal by Subject | 4
Not completed — Unable to obtain specimen | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pharmacokinetics of Daunorubicin Chemotherapy Patients
Number analyzed (Participants) | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 99
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.5 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 13
  White | 82
  More than one race | 2
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Population Estimates for Daunorubicin Hydrochloride Clearance
Description: Pharmacokinetic parameters of Daunorubicin hydrochloride will be analyzed, samples were drawn according to the following schedule: prior to the drug infusion, at the midpoint of the infusion if infusion is ≥ 30 min in duration, end of infusion and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 (when feasible) hours after the end of the infusion. Samples will also be collected at 24, 48, and 72 (when feasible) hours after the end of the infusion. The concentration time data will be analyzed by model dependent and model-independent means. Pharmacokinetic data will be analyzed using ADAPT II software (Biomedical Simulations Resource, University of Southern California). Mean Daunorubicin hydrochloride Clearance will be assessed.
Time Frame: Prior to drug infusion, midpoint, and end of infusion. Also 0.5,1,1.5,2,3,4,6,8 and 12 hours after end of infusion.
Population: There were 107 patients enrolled, 4 participants withdrew consent and there was 1 patient with insufficient specimen. 4 other participants were not analyzed as all sample time points were required for analysis and were not available.
Measure: Mean (Standard Deviation); unit: L/m2/hr
Arm/Group | Pharmacokinetics of Daunorubicin Chemotherapy Patients
Number analyzed (Participants) | 98
L/m2/hr | 116 (14)

2. Primary Outcome: Population Estimates for Daunorubicin Hydrochloride Volume of Distribution
Description: Pharmacokinetic parameters of Daunorubicin hydrochloride will be analyzed, samples were drawn according to the following schedule: prior to the drug infusion, at the midpoint of the infusion if infusion is ≥ 30 min in duration, end of infusion and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 (when feasible) hours after the end of the infusion. Samples will also be collected at 24, 48, and 72 (when feasible) hours after the end of the infusion. The concentration time data will be analyzed by model dependent and model-independent means. Pharmacokinetic data will be analyzed using ADAPT II software (Biomedical Simulations Resource, University of Southern California). Mean volume of distribution will be assessed.
Time Frame: Prior to drug infusion, midpoint, and end of infusion. Also 0.5,1,1.5,2,3,4,6,8 and 12 hours after end of infusion.
Population: There were 107 patients enrolled, 4 participants withdrew consent and there was 1 participant with insufficient specimen. 4 other participants were not analyzed as all samples time points were required for analysis and were not available.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Pharmacokinetics of Daunorubicin Chemotherapy Patients
Number analyzed (Participants) | 98
Liter | 68.1 (24)

3. Secondary Outcome: Relationship Between Body Composition and the Pharmacokinetics of Daunorubicin Hydrochloride
Description: Mean (standard deviation) of daunorubicin hydrochloride clearance will be summarized by Body composition (<30% versus >=30%)
Time Frame: Length of study
Reporting Status: Not Posted

4. Secondary Outcome: Correlation of the Pharmacokinetics of Daunorubicin Hydrochloride With Gender, Age, or Ethnic Background
Description: Mean (standard deviation) of daunorubicin hydrochloride clearance will be summarized by Gender (Male versus Female), Age group (<median age versus >=median age in years), Race (White vs. Black vs. Other)
Time Frame: Length of Study
Reporting Status: Not Posted

5. Secondary Outcome: Relationship Between Pharmacokinetics and Toxicity
Description: Mean (standard deviation) of daunorubicin hydrochloride clearance will be summarized for occurrence of various toxicities
Time Frame: Length of Study
Reporting Status: Not Posted

6. Secondary Outcome: Relationship Between Pharmacokinetics, Renal and Hepatic Function, and Complete Blood Count
Description: Mean (standard deviation) of daunorubicin hydrochloride clearance will be summarized by organ function/baseline laboratory values
Time Frame: Length of Study
Reporting Status: Not Posted

7. Secondary Outcome: Relationship Between Pharmacokinetics, and Genetic Polymorphisms
Description: Mean (standard deviation) of daunorubicin hydrochloride clearance will be summarized by genotype
Time Frame: Length of Study
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Pharmacokinetics of Daunorubicin Chemotherapy Patients
Serious Adverse Events (participants affected / at risk) | 0/107
Other Adverse Events (participants affected / at risk) | 50/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pharmacokinetics of Daunorubicin Chemotherapy Patients (N=107)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 26
White blood cell decreased (Blood and lymphatic system disorders) | 33
Lymphocyte count decreased (Blood and lymphatic system disorders) | 21
Neutrophil count decreased (Blood and lymphatic system disorders) | 30
Platelet count decreased (Blood and lymphatic system disorders) | 27
Fibrinogen (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Constipation (Metabolism and nutrition disorders) | 1
Diarrhea (Metabolism and nutrition disorders) | 2
Mucositis oral (Metabolism and nutrition disorders) | 1
Nausea (Metabolism and nutrition disorders) | 1
Proctitis (Metabolism and nutrition disorders) | 1
Vomiting (Metabolism and nutrition disorders) | 1
"Vascular disorders - Other, specify" (Vascular disorders) | 1
Enterocolitis infectious (Infections and infestations) | 1
Febrile neutropenia (Infections and infestations) | 9
"Infections and infestations - Other, specify" (Infections and infestations) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypercholestremia (Metabolism and nutrition disorders) | 1
GGT increased (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Lipase (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 1
Pain (General disorders) | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.